CLINICAL TRIAL: NCT04822831
Title: The Effect of 45 Degree Semi-recumbent Position With Upper Limb Exercise Training on Long-term Ventilator-dependent Patients
Brief Title: The Effect of Semi-recumbent Position With Exercise Training on Long-term Ventilator-dependent Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taoyuan General Hospital (Other Government)
Responsible Party: Principal Investigator, Se-Hua Lin, Head Nurse, Taoyuan General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SeHLin
Record Dates: First submitted 2021-03-23; First posted 2021-03-30 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Mechanical Ventilation; Difficult Intubation; Position; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This study used repeated experimental measurements and purpose sampling, and we invited patients in respiratory care ward (RCW) in northern Taiwan. They were randomly assigned to the experimental group and the control group. The experimental group was given 45 degree Semi-sitting for 2hrs and upper-limb exercise training 10mins once a day. The control group was just continue the routine treatment. After 4 weeks, we measure the respiratory parameters such as maximum inspiratory pressure (MIP), tidal volume (VT), minute ventilation (MV), and rapid shallow breathing index(RSBI) of these two groups, and used GEE to compare with them. To find the differences in respiratory parameters, ventilator detachment rate,
Who Masked: Participant
Masking Description: The participants involved in the clinical trial who are prevented from having knowledge of the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long-term Ventilator-dependent Patients with intervention (Experimental): 45 Degree Semi-recumbent Position With Upper Limb Exercise Training on Long-term Ventilator-dependent Patients
  Interventions: Behavioral: 45 Degree Semi-recumbent Position With Upper Limb Exercise Training
- Long-term Ventilator-dependent Patients without intervention (Experimental): There is no intervention on Long-term Ventilator-dependent Patients ,and just keep routine treatment.
  Interventions: Behavioral: no 45 Degree Semi-recumbent Position With Upper Limb Exercise Training

INTERVENTIONS:
Behavioral: 45 Degree Semi-recumbent Position With Upper Limb Exercise Training — The experimental group was given 45 degree Semi-sitting 2 hrs and upper-limb exercise training 10 mins once a day, and this intervention kept 4 weeks.
  Other Names: 45 Degree Semi-sitting Position With Upper Limb Exercise Training
  Arms: Long-term Ventilator-dependent Patients with intervention
Behavioral: no 45 Degree Semi-recumbent Position With Upper Limb Exercise Training — The control group was with usual treatment.
  Other Names: no other intervention
  Arms: Long-term Ventilator-dependent Patients without intervention

SUMMARY:
Prolonged mechanical ventilation patients rely on medical expenses per year had increased by nearly 20 billion in 15 years, so it is worthwhile to explore how to improve the respiratory function and even their quality of life of patients in Respiratory care wards (RCWs). This study used repeated experimental measurements and purpose sampling, and the investigators invited patients in respiratory care ward in northern Taiwan. They were randomly assigned to the experimental group and the control group. The experimental group was given 45 degree Semi-sitting 2 hrs and upper-limb exercise training 10 mins once a day. There were 29 prolonged mechanical ventilation (PMV) patients in the experimental group and 26 in the control group. Our conclusions showed that PMV patients can significantly improve the maximum inspiratory pressure (MIP) in the post-test while performed a 45-degree semi-sitting position with upper limb training for 4 weeks. The minute ventilation (MV) has a trend of increasing month by month in the experimental group, but it is necessary to consider whether it is due to the improvement of lung function or just cause of the increased oxygen consumption and accelerated respiratory rate, so it can not be inferred to improvement of the patient's condition or lung function.

DETAILED DESCRIPTION:
Background: Prolonged mechanical ventilation patients rely on medical expenses per year had increased by nearly 20 billion in 15 years. However, the high cost shows the high morbidity rate, high mortality rate and low ventilator weaning rate of prolonged mechanical ventilation patients, so it is worthwhile to explore how to improve the respiratory function and even their quality of life of patients in the respiratory care ward (RCW).

OBJECTIVE: To investigate the improvement of respiratory function and the effect of respirator detachment in 45-degree semi-sitting and upper limb training, and to understand the correlation between this training activity and death risk.

METHODS: This study used repeated experimental measurements and purpose sampling, and the investigators invited patients in the respiratory care ward (RCW) in northern Taiwan. They were randomly assigned to the experimental group and the control group. The experimental group was given 45 degree Semi-sitting 2hrs and upper-limb exercise training 10mins once a day. After 4 weeks, the investigators measure the respiratory parameters such as the maximum inspiratory pressure (MIP), the tidal volume (VT), the minute ventilation (MV), and the rapid shallow breathing index(RSBI) of these two groups, and used the generalized estimating equation (GEE) to compare with them.

ELIGIBILITY:
Inclusion Criteria

* respiratory care ward (RCW) cases using mechanical ventilators
* 20 years old ≦ age ≦ 89 years old
* Those who used antibiotics without infection and fever (body temperature >38.5℃) in the past 3 days
* the fraction of inspiration O2(FiO2)≦50% and the positive end expiratory pressure(PEEP)≦10
* 90 mm-Hg≦ systolic blood pressure(SBP) ≦160 mm-Hg
* 60 beats/min≦ heart rate(HR) ≦130 beats/min without arrhythmia
* 12 times/min≦ respiratory rate(RR) ≦35 times/min
* 90%≦ oxygen saturation by pulse oximetry (SPO2) ≦100%
* Patients with spontaneous breathing
* Digestible without continuous feeder

Exclusion Criteria:

* respiratory care ward (RCW) cases without mechanical ventilators
* Age <20 years old or age>89 years old
* Those who have been infected with fever in the past 3 days (body temperature >38.5℃) and are taking antibiotic
* the fraction of inspiration O2(FiO2) >50% and the positive end expiratory pressure(PEEP)>10
* systolic blood pressure(SBP)< 90 mm-Hg or systolic blood pressure(SBP) >160 mm-Hg
* heart rate(HR)<60 beats/min or heart rate(HR)>130 beats/min and arrhythmia
* respiratory rate(RR)<12 times/minute or respiratory rate(RR)>35 times/minute
* oxygen saturation by pulse oximetry (SPO2) <90%
* Patients without spontaneous breathing
* Poor digestion and use of continuous feeders

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
maximum inspiratory pressure (MIP) | Change from maximum inspiratory pressure (MIP) at 1 month
  After doing intervention for 4 weeks, we measure the maximum inspiratory pressure (MIP) of these two groups
tidal volume (VT) | Change from tidal volume (VT) at 1 month
  After doing intervention for 4 weeks, we measure the tidal volume (VT) of these two groups
minute ventilation (MV) | Change from minute ventilation (MV) at 1 month
  After doing intervention for 4 weeks, we measure the minute ventilation (MV) of these two groups
rapid shallow breathing index (RSBI) | Change from rapid shallow breathing index (RSBI) at 1 month
  After doing intervention for 4 weeks, we measure the rapid shallow breathing index (RSBI) of these two groups

CONTACTS AND LOCATIONS:
Overall Officials: Se-Hua Lin, master, Principal Investigator — Taoyuan Armed Forces General Hospital
Locations (1):
- Se-Hua Lin, Taoyuan District, Longtan Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No
we don't plan to make individual participant data (IPD) ,because the database belonged to patients and hospitals